CLINICAL TRIAL: NCT00005600
Title: Optimum Drainage of the Axilla After Lymph Node Dissection: A Randomized Prospective Study
Brief Title: Axillary Drainage Following Lymph Node Dissection in Women With Stage I or Stage II Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000067713; RMNHS-1489; EU-20004
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2005-12

CONDITIONS: Breast Cancer; Lymphedema; Perioperative/Postoperative Complications
Keywords: stage I breast cancer; stage II breast cancer; lymphedema; perioperative/postoperative complications
MeSH Terms: conditions — Breast Neoplasms; Lymphedema; Postoperative Complications

INTERVENTIONS:
Procedure: management of therapy complications

SUMMARY:
RATIONALE: The use of axillary drains may help to prevent complications following axillary lymph node dissection.

PURPOSE: This randomized clinical trial is comparing three methods of axillary drainage to see how well they work following lymph node dissection in women with stage I or stage II breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare high vacuum drainage vs low vacuum drainage vs simple tube drainage in patients undergoing axillary surgery for stage I or II breast cancer.

OUTLINE: This is a randomized study.

Patients undergo axillary dissection, then are randomized to one of three axillary drainage systems.

* Arm I: Patients receive high vacuum drainage.
* Arm II: Patients receive low vacuum drainage.
* Arm III: Patients receive simple tube drainage (no vacuum). All drains are removed when daily volumes are below 30 mL or at 5 days after surgery, regardless of drain volume.

Patients are followed at day 10 and at 3 months.

PROJECTED ACCRUAL: A total of 200 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of resectable stage I or II breast cancer
* Planned primary surgery of level II or III axillary dissection in association with one of the following:

  * Wide local excision (may be done through separate incision)
  * No breast surgery
  * Bilateral surgery allowed
* No prior mastectomy
* No immediate breast reconstruction using implants, latissimus dorsi, or rectus abdominus myocutaneous flaps at primary operation
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* See Disease Characteristics
* No prior axillary surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-11

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Gui, MD, MS, FRCS(Edin), FRCS(Eng), Study Chair — Royal Marsden NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Royal Marsden NHS Foundation Trust - London, London, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England